CLINICAL TRIAL: NCT03080597
Title: PrEP for HBCUs (Study 2)
Acronym: PrEP for HBCUs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Intelligent Automation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00076107
Record Dates: First submitted 2017-01-17; First posted 2017-03-15 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-03

CONDITIONS: At Risk for HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smartphone app condition (Experimental): English-speaking males, between the ages of 18-30, who are enrolled at a HBCU or identify as Black/African American, who are currently prescribed PrEP (Truvada) for HIV Prevention, and owners of either an Android or iOS smartphone, will be asked to use an application on their smart phones called "PrEP Smart".
  Interventions: Device: PrEP Smart app

INTERVENTIONS:
Device: PrEP Smart app — English-speaking males, between the ages of 18-30, who are enrolled at a HBCU or identify as Black/African American, who are currently prescribed PrEP (Truvada) for HIV Prevention, and owners of either an Android or iOS smartphone, will be asked to use an application on their smart phones called "PrEP Smart".an application on their smart phones called "PrEP Smart".

SUMMARY:
The investigators' overall goals are to target (a) pre-exposure prophylaxis (PrEP) uptake by addressing access and acceptability and (b) PrEP adherence among Historically Black Colleges and Universities (HBCU) students.

DETAILED DESCRIPTION:
The following is only pertaining to study 2, HBCUs. PrEP Smart (study 1) is not included in this record.

The investigators' overall goals are to target (a) pre-exposure prophylaxis (PrEP) uptake by addressing access and acceptability and (b) PrEP adherence among Historically Black Colleges and Universities (HBCU) students.

Aim 1/Study 1. Investigate uptake of PrEP services on HBCU campuses. Making PrEP available on HBCU campuses may address uptake by increasing (a) accessibility by allowing students to gain access to tenofovir disproxil fumarate/emtricitabine (TDF/FTC) without having to leave campus and (b) acceptability by providing trained practitioners and student advocates on campus to educate students on the benefits of PrEP. Aim 1a will target PrEP uptake at HBCUs at the healthcare systems level. The investigators will identify Student health centers (SHC) practitioners on 6 HBCUs (North Carolina Central, St. Augustine's, Fayetteville State University, Shaw, North Carolina A&T, and Bennett College). After a comprehensive SHC needs assessment, the investigators will train practitioners on eligibility for PrEP, pre-initiation counseling, and prescribing in partnership with the North Carolina AIDS Education and Training Center (NC AETC). The investigators will also engage key student organizations on campus and train motivated student advocates for the dissemination of information about PrEP on campus. Aim 1b will target PrEP uptake at the individual level. First, the investigators will collect data on all clinical encounters for PrEP at participating SHCs during the study period. Data will be collected on the basic demographics and risk factors necessitating the initiation of PrEP. The investigators will also collect data on PrEP initiations, as well as the number of prescriptions written in follow up during the period of study. To better understand PrEP behaviors on campus, the investigators will ask students initiated on PrEP to take a brief, anonymous questionnaire on relevant topics including: (1) PrEP awareness, (2) Motivation for initiating PrEP, (3) Perceived stigma of HIV and HIV associated risk factors on campus, and (4) Perceptions of confidentiality regarding seeking PrEP services on campus. The investigators anticipate enrolling approximately 250 students for this portion of the study.

Aim 2/Study 2. Adapt a smartphone-based contingency management (CM) application ("app") intervention designed to improve PrEP adherence. CM is a behavioral intervention that involves the systematic use of reinforcement dependent on the occurrence of a predefined behavior. CM improves adherence to antiretroviral therapy (ART) and post-exposure prophylaxis (PEP), and is currently being developed by the investigative team for PrEP. Since the cost of traditional CM interventions may be prohibitive in practice, the investigators will adapt this intervention using a lower cost reinforcement procedure and therefore improve the scalability of this adherence intervention. In a sample of young men who have sex with men (YMSM) prescribed PrEP (n = 20) over an 8 week period, Aim 2a will assess app interaction to address feasibility, Aim 2b will assess acceptability via self-report quantitative ratings and qualitative interviewing, Aim 2c will assess the validity of daily camera-based medication ingestion assessment via the app to validate medication adherence against blood tests to detect PrEP, and Aim 2d will assess barriers to adherence via app-based daily assessments following missed doses.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled as a student in a Historically Black College or University, OR identify as Black/African American
* Male
* Self-report having sex with men in the past 6 months
* 18-30 years of age
* English-speaking
* Currently prescribed PrEP (Truvada) for HIV prevention
* Participant has an Android (using v5.x.x or lollipop) or iOS (v6.0) smartphone

Exclusion Criteria:

* History of a chronic/significant medical or psychiatric condition that will interfere with study participation
* Unable to attend sessions

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by the number of times per day that subjects initiate an interaction with PrEP Smart | 8 weeks
  As measured by the number of times per day that subjects initiate an interaction with PrEP Smart
Feasibility as measured by the number of times per day that subjects respond to a PrEP Smart prompt | 8 weeks
  As measured by the number of times per day that subjects respond to a PrEP Smart prompt

SECONDARY OUTCOMES:
Acceptability will be assessed during the final laboratory visit with an open ended qualitative interview assessing overall feedback | 8 weeks
  Will be assessed during the final laboratory visit with an open ended qualitative interview assessing overall feedback.
Acceptability will be assessed by feedback specific to each of the six individual PrEP Smart features | 8 weeks
  Will be assessed by feedback specific to each of the six individual PrEP Smart features.
Adherence will be assessed by the number of times that PrEP was taken daily over the 8 week period and the number of times that it was taken outside of a one hour window in which it was prescribed | 8 weeks
  Will be assessed by the number of times that PrEP was taken daily over the 8 week period and the number of times that it was taken outside of a one hour window in which it was prescribed.

CONTACTS AND LOCATIONS:
Overall Officials: John T Mitchell, Ph.D., Principal Investigator — Study Principal Investigator
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided